CLINICAL TRIAL: NCT06359782
Title: A Phase II Trial on the Safety and Efficacy of C1 Inhibitor for the Acute Management of Subarachnoid Hemorrhage
Brief Title: Complement Inhibition: Attacking the Overshooting Inflammation @Fter Subarachnoid Hemorrhage (CIAO@SAH)
Acronym: CIAO@SAH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haaglanden Medical Centre (Other)
Collaborators: Leiden University Medical Center (Other); Takeda (Industry)
Responsible Party: Principal Investigator, Wouter Moojen, Principal Investigator, Haaglanden Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL76082.058.20
Record Dates: First submitted 2024-03-22; First posted 2024-04-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Complement C1 Inhibitor Protein; SERPING1 protein, human

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized, double-blind, placebo-controlled, phase II trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- C1-esterase inhibitor (Cinryze) (Experimental): One group receiving study medication (C1-esterase inhibitor Cinryze)
  Interventions: Drug: C1 Esterase Inhibitor Injection [Cinryze]
- Placebo (Placebo Comparator): One group receiving placebo medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C1 Esterase Inhibitor Injection [Cinryze] — C1 Esterase Inhibitor Injection [Cinryze]
  Other Names: Cinryze
  Arms: C1-esterase inhibitor (Cinryze)
Drug: Placebo — Sodium Chloride /physiological saline (0.9%) in equal volume dosed intravenous
  Arms: Placebo

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) can lead to devastating outcomes for patients, like cognitive decline. This is caused by early brain injury (EBI) followed by delayed cerebral ischemia (DCI). Neuroinflammation, triggered by the complement system, has been investigated to be a key mediator in the pathophysiology of EBI and DCI. Inhibition of the complement system is therefore considered to be a potentially important new treatment for SAH.

This trial aims to study the safety and efficacy of C1-inhibitor Cinryze, an approved inhibitor of the complement system, compared to placebo in patients with SAH. By temporarily blocking the complement system we hypothesize limitation of delayed cerebral ischemia and a more favourable clinical outcome for SAH patients due to a decrease in the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of aneurysmal subarachnoid hemorrhage on CT-scan;
* Age ≥ 18 years on admission;
* WFNS grade 1-5.

Exclusion Criteria:

* Subarachnoid hemorrhage deemed most likely of 'peri mesencephalic' origin after consideration of history, clinical examination and radiological findings (including angiographic imaging); (not originated from an aneurysm and patients have by definition a favourable clinical outcome)
* Subarachnoid hemorrhage deemed most likely of post-traumatic origin after consideration of history, clinical examination and radiological findings (including angiographic imaging); (does not occur spontaneous)
* Participation in another clinical therapeutic study;
* Patients with definite infaust prognosis on arrival and/or expected death within 24 hours of admission
* Patients with a known hereditary complement deficiency (including hereditary angioedema);
* Patients with a history of sensibility to blood products or C1-inhibitor;
* Patients with a history of thrombosis (when known at time of inclusion);
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delayed cerebral ischemia (DCI) | To be determined between day 4 and day 14 of admission
  Defined as either a new focal neurological impairment, or a decrease of at least 2 points on the Glasgow Coma Scale. This should last for at least 1 hour, is not apparent immediately after aneurysm occlusion, and cannot be attributed to other causes by means of clinical assessment, CT or MRI scanning of the brain, and appropriate laboratory studies.
Number of participants with complications during hospitalization. | Up to 1 year after admission
  Complication rate during hospitalization

SECONDARY OUTCOMES:
Number of participants with cerebral infarction on brain CT | at 14 days after admission
Number of participants dying | Up to 1 year after admission
  Mortality rate
Neurological condition measured by Glasgow Coma Scale | During the first 14 days
  Measured daily, minimum value of 3, maximal value of 15, higher scores mean a better outcome
Complement activity markers measured in serum and CSF | Before IV administration of C1-INH or placebo, and after 48 hours and 96 hours after IV administration
  WIESLAB, C3b/C, C4b/C, C5b-9 ELISA assays, CH50/AC50
Inflammatory markers measured in serum and CSF | Before IV administration of C1-INH or placebo, and after 48 hours and 96 hours after IV administration
  TNF-alpha, intraleukins
Number of days in the hospital | Up to 1 year
  Hospital length of stay
Number of ICU days | Up to 1 year
  ICU length of stay
Number of ventilator days | Up to 1 year
  Ventilator days
Clinical outcome | At 6 months
  Modified Ranking Scale, minimum value 0, maximum value 6, higher score means worse outcome
Clinical outcome | At 6 months
  Glasgow Outcome Scale Extended, minimum value 1, maximum value 8, higher score means better outcome
Clinical outcome | At 6 months
  Barthel Index, minimum value 0, maximum value 100, higher score means better outcome
Clinical outcome | At 6 months
  Montreal Cognitive assessment, minimum value 0, maximum value 30, higher score means better outcome
Clinical outcome | At 6 months
  Quality of Life (EQ-5D-5l), minimum value -0.51, maximum value 1, higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Moojen, MD PHD, Principal Investigator — Haaglanden Medisch Centrum
Locations (1):
- Haaglanden Medical Centre, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No